CLINICAL TRIAL: NCT02704897
Title: Can a Smartphone-delivered Tool Facilitate the Assessment of Surgical Site Infection, and Result in Earlier Treatment? A Randomized-controlled Trial in Emergency Surgery Patients.
Brief Title: Tracking Wound Infection With Smartphone Technology
Acronym: TWIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AC16032
Record Dates: First submitted 2016-03-02; First posted 2016-03-10 (Estimated); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Arm (Experimental): Wound assessment tool - delivered via a smartphone. A link will be sent to participants on discharge, which can be accessed at any point should they have concerns about their wound.
  They will also be sent the tool at 3 additional time-points.
  Interventions: Other: Wound Assessment Tool
- Control Arm (No Intervention): Normal Post-operative Care

INTERVENTIONS:
Other: Wound Assessment Tool — A set of questions relating to the symptoms of wound infection
  Arms: Intervention Arm

SUMMARY:
This study aims to evaluate if a smartphone-delivered tool can help assess for wound infections, and if this improves access to care and results in earlier treatment. Participants will be randomised to one of two groups. The intervention group will receive the smartphone-delivered wound assessment tool (SWAT), to access if they have concerns about their wound. The trial period is 30 days.

DETAILED DESCRIPTION:
Surgical site infection (SSI) is defined by the Centre for Disease Control and Prevention (CDC) as an infection in the skin and soft tissues of a surgical wound, within 30 days of the operation. It is a common problem, and complicates 2-10% of general surgery operations. The majority of cases are diagnosed outside of hospital and can be treated with oral antibiotics.

Interest in the use of technology in medicine is increasing, with the potential that more advanced technology will help facilitate communication between clinicians and patients, aid in the assessment of patients, and improve clinical decision making. Over two-thirds of people now own smartphones, and regularly use them to access the internet. The investigators wish to use a smartphone delivered questionnaire to help assess SSI and see if this improves access to care and time to treatment.

The investigators will be recruiting emergency surgery patients with smartphones at the Royal Infirmary and Western General Hospitals in Edinburgh.

Participants will be divided into two groups. One group will receive the wound assessment tool, if they are concerned about their wound, they can use the tool to answer a series of questions. If their answers suggest SSI, a clinician will contact them to advise further assessment and treatment. The participants will also be asked to respond to the tool three times during the trial (to collect responses from those without symptoms), and upload photos of their wounds to a secure database.

The second group of participants will receive normal post-operative care.

After 30 days, participants will have a follow-up consultation, to determine if they have had a wound infection (this can be via telephone or face-to-face, according to participant preference). They will also answer questions about their experience of the study, and use of services.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Abdominal Surgery Patients
* Smartphone Owners
* Able to give valid consent

Exclusion Criteria:

* Significant visual impairment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Time from surgery to treatment for surgical site infection | Outcome assessed at 30 day follow-up
  Measured in days from surgery to commencing antibiotic treatment

SECONDARY OUTCOMES:
Service Usage | Assessed at 30 day follow-up
  Number of attendances at General Practice (GP) and Accident and Emergency (A&E).
Access to Services | Assessed at 30 day follow-up
  How long in days between experiencing first symptom and being reviewed by A&E, GP or surgical team

CONTACTS AND LOCATIONS:
Overall Officials: Ewen Harrison, BM CHB, Principal Investigator — University of Edinburgh
Locations (2):
- United Kingdom (2):
  - Royal Infirmary Edinburgh, Edinburgh
  - Western General Hospital, Edinburgh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McLean KA, Mountain KE, Shaw CA, Drake TM, Ots R, Knight SR, Fairfield CJ, Sgro A, Skipworth RJE, Wigmore SJ, Potter MA, Harrison EM. Can a smartphone-delivered tool facilitate the assessment of surgical site infection and result in earlier treatment? Tracking wound infection with smartphone technology (TWIST): protocol for a randomised controlled trial in emergency surgery patients. BMJ Open. 2019 Oct 3;9(10):e029620. doi: 10.1136/bmjopen-2019-029620. PMID 31585971
- See also: Public Health England. Surgical site infection surveillance service (SSISS). (2014). — https://www.gov.uk/guidance/surgical-site-infection-surveillance-service-ssiss
- See also: CDC/OID/NCEZID/DHQP. 9 surgical site infection (SSI) event. (2016). — http://www.cdc.gov/nhsn/PDFs/pscManual/9pscSSIcurrent.pdf